CLINICAL TRIAL: NCT05010005
Title: Phase I Multicenter Study of Ruxolitinib and Duvelisib in Relapsed or Refractory T- or NK-Cell Lymphomas
Brief Title: A Study of Ruxolitinib and Duvelisib in People With Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-176
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: T-cell Lymphomas; NK-Cell Lymphomas; T-cell Prolymphocytic Leukemia; T-cell Large Granular Lymphocyte Leukemia
Keywords: mature T-cell lymphomas; Ruxolitinib; Duvelisib; Relapsed or Refractory; 21-176; T-cell Large Granular Lymphocyte Leukemia; T-cell Prolymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, Prolymphocytic, T-Cell; Leukemia, Large Granular Lymphocytic; Recurrence | interventions — ruxolitinib; duvelisib

STUDY DESIGN:
Intervention Model Description: This phase I study includes a dose escalation phase and a dose expansion phase.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib and Duvelisib (Experimental): Ruxolitinib 20mg BID plus Duvelisib 25mg, 50mg, or 75mg BID. Patients will be instructed to take duvelisib and ruxolitinib by mouth every 12 hours, the same time each day, +/- 2 hours. Duvelisib and ruxolitinib will be provided via the institutional investigational pharmacy. The researchers will utilize a dose-escalation standard 3+3 design in which we evaluate 3 doses of duvelisib (25mg BID, 50mg BID, and 75mg BID) in combination with ruxolitinib 20mg BID. A minus-1 dose level of duvelisib (15mg BID) can be used if de-escalation is needed. The cohort expansion phase will have two treatment groups JAK/STAT activation or mutation present or JAK/STAT activation or mutation absent or unknown. Upon discussion with PI, the treating physician may increase dose up to 20 mg of ruxotlinib and/or 25 mg of duvelisib when deemed clinically favorable. T-prolymphocytic leukemia (T-PLL) and T-follicular helper (TFH) lymphoma expansion: Further expansion for patients with T-PLL and TFH lymphomas.
  Interventions: Drug: Ruxolitinib; Drug: Duvelisib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 20mg BID
Drug: Duvelisib — Duvelisib 25mg, 50mg, or 75mg BID

SUMMARY:
This study will test the safety of ruxolitinib, given at one dose that does not change, and duvelisib, given at different doses, to find out what effects, if any, the study treatment has on people with relapsed or refractory NK-cell or T-cell lymphoma.

This study has three parts: dose escalation (Part 1), dose expansion (Part 2), and TFH/T-PLL cohort expansion (Part 3).

ELIGIBILITY:
Inclusion Criteria:

a) Pathologically-confirmed mature T-cell lymphomas at the enrolling institution.

Permitted histologies include (for dose escalation and expansion):

i) Stage ≥Ib CTCL, which has relapsed or progressed after at least two systemic therapies. In order to ensure balanced enrollment for patients with systemic T-cell lymphoma and CTCL, a maximum of 15 CTCL patients will be enrolled in expansion cohort.

ii) Systemic anaplastic large cell lymphoma that has relapsed after therapy containing brentuximab vedotin.

iii) T-cell prolymphocytic leukemia (treatment naïve permitted)

For the following histologies, patients are required to have received at least 1 prior therapy (dose escalation and expansion):

iv) T-cell large granular lymphocytic leukemia

v) Aggressive NK-cell leukemia

vi) Adult T-cell leukemia/lymphoma

vii) Extranodal NK/T- cell lymphoma, nasal type

viii) Enteropathy-associated T-cell lymphoma

ix) Monomorphic epitheliotropic intestinal t-cell lymphoma

x) Hepatosplenic T cell lymphoma

xi) Subcutaneous panniculitis-like T-cell lymphoma

xii) Primary cutaneous anaplastic large cell lymphoma

xiii) Primary cutaneous gamma/delta T-cell lymphoma

xiv) Primary cutaneous CD8-positive aggressive epidermotropic cytotoxic T-cell lymphoma

xv) Peripheral T-cell lymphoma, not otherwise specified

xvi) Angioimmunoblastic T cell lymphoma

xvii) Follicular T-cell lymphoma

xviii) Nodal peripheral T-cell lymphoma wih T follicular helper phenotype

b) Nodal periphal T-cell lymphoma wih T follicular helper phenotype Specific for T-PLL and TFH lymphoma expansion: histologies must be pathologically confirmed at the enrolling institutions i) T-cell prolymphocytic leukemia (treatment naïve permitted) ii) T-follicular helper lymphomas (must have received at least 1 prior treatment)

c) Age ≥18 years at time of enrollment

d) Performance status, as assessed in the ECOG grading system, ≤2

e) Laboratory criteria.

Laboratory criteria

i) For dose escalation phase:

1. Absolute neutrophil count ≥1.0 K/mcL (Note: growth factor is allowed)
2. Platelet count ≥80 K/μl or ≥50 K/μl if due to lymphoma
3. Creatinine ≤1.5 × ULN OR Measured calculated creatinine clearance ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN

i. Creatinine clearance should be calculated per institutional standard

d. Direct bilirubin ≤1.5x upper limit of normal (ULN) or ≤3x ULN if documented hepatic involvement with lymphoma, or ≤5x ULN if history of Gilbert's syndrome; AST and ALT ≤ 3x ULN; or ≤ 5x ULN if due to lymphoma involvement

ii) For dose expansion phase and T-PLL/TFH lymphoma expansion:

1. Absolute neutrophil count ≥1.0 K/mcL or ≥0.5 K/mcL if due to lymphoma or ≥0.0 K/mcL if due to T-PLL or large granular lymphocytic leukemia (LGL) (Note: growth factor is allowed).
2. Platelet count ≥80 K/μl or ≥50 K/μl if due to lymphoma
3. c. Creatinine ≤1.5 × ULN OR Measured calculated creatinine clearance ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN

i. Creatinine clearance should be calculated per institutional standard d. Direct bilirubin ≤1.5x upper limit of normal (ULN) or ≤3x ULN if documented hepatic involvement with lymphoma, or ≤5x ULN if history of Gilbert's syndrome; AST and ALT ≤ 3x ULN; or ≤ 5x ULN if due to lymphoma involvement

f) Measurable disease, defined by at least one of the following:

* Revised International Working Group Classification for systemic lymphoma19
* Atypical T lymphocytes quantifiable by flow cytometry or morphology in the peripheral blood or bone marrow
* mSWAT (Modified Severity Weighted Assessment Tool) >0

  g) Ability to swallow pills

  h) Women of reproductive potential* must have a negative serum or urine β human chorionic gonadotropin (βhCG) pregnancy test within 14 days of initiating therapy. All women of reproductive potential and all sexually active male patients must agree to use adequate methods of birth control (e.g. latex condoms) throughout the study and for 3 months after the last dose of study drug.
  * A woman of reproductive potential is a sexually-mature woman who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months).
* The effects of duvelisib on conception, pregnancy, and lactation are unknown. Since duvelisib has not been evaluated in pregnant or nursing women, the treatment of pregnant women or women of childbearing potential who are not using a highly effective contraception is contraindicated.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant women. (Lactating women must agree not to breast feed while taking study medications).
3. Prior allogeneic stem cell transplant within 6 months of starting treatment or patients with active GVHD requiring immunosuppression.

a. Prior allogeneic stem cell transplant may be allowed after discussion with MSK PI if no GVHD or immunosuppression is present at time of enrollment...

d) Prior use of duvelisib or ruxolitinib if either agent was discontinued due to toxicity.

e) Previous systemic anti-cancer therapy for TCL within 14 days of initiating study drug

a. Patients who have received localized RT as part of their immediate prior therapy may be allowed to enroll with shorter washout period after discussion with the MSK Principal Investigator.

i. Patients receiving treatment with single agent ruxolitinib or duvelisib may be allowed to enroll onto the study without a washout period

b. Systemic corticosteroids must be tapered to 20mg/day or less prednisone (or equivalent) upon start of investigational treatment.

c. Topical steroids for CTCL is permitted on study.

f) Ongoing use of immunosuppressant medications, including corticosteroids greater than 20mg of prednisone or equivalent at the time of enrollment

g) History of chronic liver disease, veno-occlusive disease, or current alcohol abuse

h) Administration of a live vaccine within 6 weeks of first dose of study drug.

i) Prior surgery or gastrointestinal condition that may adversely affect drug absorption (e.g., gastric bypass surgery, gastrectomy)

j) Patients with HIV infection if they meet either of the below criteria:

i. detectable viral load ii. undetectable viral load with CD4 count <200 or not taking anti-retroviral medications.

k) Patients with chronic hepatitis B or C as defined by positive hepatitis B or C serology:

* Subjects with a negative HBsAg and a positive HBcAb require an undetectable/negative hepatitis B DNA test (e.g., polymerase chain reaction [PCR] test) to be enrolled, and must receive hepatitis B prophylaxis until at least 6 months after completion of study drug(s).

  l) Subjects with active CMV (defined as positive CMV PCR with clinical manifestations consistent with active CMV infection) and requiring therapy. Carriers will be monitored per institutional guidelines.

  m) Unable or unwilling to receive prophylaxis against pneumocystis, herpes simplex virus, or herpes zoster

  g) Use of medications or consumption of foods that are strong inducers or inhibitors of CYP3A
* Such agents must be discontinued at least 2 weeks prior to study intervention
* Patients who (after enrollment) require use of a strong CYP3A4 inhibitor to treat a fungal/mold infection will require dose reductions n) Receipt of treatment for tuberculosis within 2 years prior to enrollment

  o) Receiving therapy for another primary malignancy (other than T-cell lymphoma).
* Patients with more than one type of lymphoma may be enrolled after discussion with the MSK Principal Investigator.
* Early-stage cutaneous basal cell and squamous cell carcinomas are permissible
* Adjuvant or maintenance therapy to reduce the risk of recurrence of other malignancy is potentially permissible after discussion with the MSK Principal Investigator.

  p) Known central nervous system or meningeal involvement by TCL (in the absence of symptoms, investigation into central nervous system involvement is not required).

  q) Unstable or severe uncontrolled medical condition (e.g., unstable cardiac function, unstable pulmonary condition) or any important medical illness that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Assessment for MTD/optimal dose | 1 year
  3 subjects will be enrolled and followed for eight weeks of safety assessments. If no DLT is observed after all three subjects have been observed for eight weeks, a second cohort of 3 subjects will be enrolled at the next highest dose level. Cohorts will continue to be enrolled and observed until one subject experiences a DLT or the maximum dose level is reached with 0 or 1/6 DLTs.

SECONDARY OUTCOMES:
Estimate the disease control rate | 6 months
  combined complete response, partial response, and stable disease for 6 months with improvement in cytopenia
Estimate the disease control rate (R+D in patients with T-PLL and TFH lymphomas) | 6 months
  combined complete response and partial response , and stable disease for 6 months with improvement in cytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of Miami (Data Collection Only), Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/